CLINICAL TRIAL: NCT01689753
Title: Prevention of Tunneled Cuffed Hemodialysis Catheter-Related Dysfunction and Bacteremia by the TEGO® Connector: A Single-Center Randomized Controlled Trial
Brief Title: Effect of the TEGO Connector in Preventing Tunneled Cuffed Hemodialysis Catheters From Dysfunction and/or Bacteremia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Joëlle Nortier, MD, PhD, MD, PhD, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P2009/021
Record Dates: First submitted 2012-07-23; First posted 2012-09-21 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Other Complication of Vascular Dialysis Catheter
Keywords: Renal dialyse; Catheter, indwelling; Catheter-related infection
MeSH Terms: conditions — Catheter-Related Infections | interventions — trisodium citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TEGO® connector (Experimental): The TEGO® connector is used during 3 consecutive hemodialyse. After each dialysis session, the dead space of the catheter is flushed with NaCl 0.9%.
  Interventions: Device: TEGO connector®
- Trisodium citrate (Active Comparator): After each dialysis, the dead space of the catheter is filled with trisodium citrate 46.7% (Citralock®).
  Interventions: Drug: Trisodium citrate

INTERVENTIONS:
Device: TEGO connector®
  Arms: TEGO® connector
Drug: Trisodium citrate
  Other Names: Citralock®
  Arms: Trisodium citrate

SUMMARY:
The aim of the trial was to assess whether use of the TEGO connector was able to reduce the incidence of a composite endpoint of TCC-related dysfunction (TCC-D)or TCC-related bacteremia (TCC-B) in chronic hemodialysis (HD) patients carrying the TEGO® connector vs controls receiving trisodium citrate 46.7%.

DETAILED DESCRIPTION:
The TEGO® connector (ICU Medical, www.icumed.com) is a closed positive pressure system, flushed with 0.9% sodium chloride and attached on the hubs of the TCC. As recommended by the producer, the TEGO® remains during 3 consecutive HD sessions and is changed every week. By constituting a mechanical barrier, it could be an interesting alternative to reduce the intraluminal contamination and the risk of TCC-B.

The TEGO® connector is supposed to provide an automatic positive displacement of fluid at the end of each TCC flush. This positive pressure could prevent the reflux of blood into the TCC lumen, possibly resulting in TCC-D.

As the impact of the TEGO® connector on TCC-D and TCC-B has never been studied, we conducted a randomized controlled study in our center by comparing the anti-thrombotic and anti-infectious efficacy of the TEGO® connector to trisodium citrate 46.7% (Citralock®, Dirinco, www.citra-lock.com) . The global cost of both procedures was also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult HD patients, prevalent or incident,carrying a tunneled cuffed catheter
* Tunneled cuffed catheter providing a mean blood flow superior to 250 ml/min
* Patients having signed an informed consent

Exclusion Criteria:

* Mature arterio-venous fistula
* Episode of TCC-related bacteremia 1 week before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Incidence rate of tunneled cuffed catheter-related dysfunction or bacteremia (composite endpoint) | 16 months
  Tunneled cuffed catheter dysfunction was defined by the requirement of urokinase and/or a mean blood flow < 250 ml/min during two consecutive hemodialysis sessions. Tunneled cuffed catheter bacteremia was defined by ≥ 2 positive qualitative and/or quantitative positive blood cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Joëlle Nortier, MD, PhD, Principal Investigator — Nephrology Dept, Erasme Hospital. Université Libre de Bruxelles, Brussel
Locations (1):
- Erasme Hospital, Anderlecht, Brussels Capital, Belgium

REFERENCES:
- [Result] Vascular Access 2006 Work Group. Clinical practice guidelines for vascular access. Am J Kidney Dis. 2006 Jul;48 Suppl 1:S176-247. doi: 10.1053/j.ajkd.2006.04.029. No abstract available. PMID 16813989
- [Result] Di Iorio BR, Bellizzi V, Cillo N, Cirillo M, Avella F, Andreucci VE, De Santo NG. Vascular access for hemodialysis: the impact on morbidity and mortality. J Nephrol. 2004 Jan-Feb;17(1):19-25. PMID 15151255
- [Result] Weijmer MC, van den Dorpel MA, Van de Ven PJ, ter Wee PM, van Geelen JA, Groeneveld JO, van Jaarsveld BC, Koopmans MG, le Poole CY, Schrander-Van der Meer AM, Siegert CE, Stas KJ; CITRATE Study Group. Randomized, clinical trial comparison of trisodium citrate 30% and heparin as catheter-locking solution in hemodialysis patients. J Am Soc Nephrol. 2005 Sep;16(9):2769-77. doi: 10.1681/ASN.2004100870. Epub 2005 Jul 20. PMID 16033861
- [Result] Weijmer MC, Debets-Ossenkopp YJ, Van De Vondervoort FJ, ter Wee PM. Superior antimicrobial activity of trisodium citrate over heparin for catheter locking. Nephrol Dial Transplant. 2002 Dec;17(12):2189-95. doi: 10.1093/ndt/17.12.2189. PMID 12454232
- [Result] Eloot S, De Vos JY, Hombrouckx R, Verdonck P. How much is catheter flow influenced by the use of closed luer lock access devices? Nephrol Dial Transplant. 2007 Oct;22(10):3061-4. doi: 10.1093/ndt/gfm314. Epub 2007 Jun 27. PMID 17597088
- [Result] Bosma JW, Siegert CE, Peerbooms PG, Weijmer MC. Reduction of biofilm formation with trisodium citrate in haemodialysis catheters: a randomized controlled trial. Nephrol Dial Transplant. 2010 Apr;25(4):1213-7. doi: 10.1093/ndt/gfp651. Epub 2009 Nov 30. PMID 19948873
- [Result] Shanks RM, Sargent JL, Martinez RM, Graber ML, O'Toole GA. Catheter lock solutions influence staphylococcal biofilm formation on abiotic surfaces. Nephrol Dial Transplant. 2006 Aug;21(8):2247-55. doi: 10.1093/ndt/gfl170. Epub 2006 Apr 20. PMID 16627606
- [Result] Punt CD, Boer WE. Cardiac arrest following injection of concentrated trisodium citrate. Clin Nephrol. 2008 Apr;69(4):317-8. doi: 10.5414/cnp69317. No abstract available. PMID 18397711
- [Result] Power A, Duncan N, Singh SK, Brown W, Dalby E, Edwards C, Lynch K, Prout V, Cairns T, Griffith M, McLean A, Palmer A, Taube D. Sodium citrate versus heparin catheter locks for cuffed central venous catheters: a single-center randomized controlled trial. Am J Kidney Dis. 2009 Jun;53(6):1034-41. doi: 10.1053/j.ajkd.2009.01.259. Epub 2009 Apr 25. PMID 19394731
- [Derived] Bonkain F, Racape J, Goncalvez I, Moerman M, Denis O, Gammar N, Gastaldello K, Nortier JL. Prevention of tunneled cuffed hemodialysis catheter-related dysfunction and bacteremia by a neutral-valve closed-system connector: a single-center randomized controlled trial. Am J Kidney Dis. 2013 Mar;61(3):459-65. doi: 10.1053/j.ajkd.2012.10.014. Epub 2012 Dec 8. PMID 23228946